CLINICAL TRIAL: NCT07223008
Title: A Pilot Study of Safety and Feasibility of Bilateral Middle Meningeal Artery Embolization (bMMAE) in Patients With Refractory Chronic Migraine Headache: The MMAE-MIGRAINE Trial
Brief Title: Bilateral Embolization of the Middle Meningeal Arteries for Refractory Chronic Migraine
Acronym: MMAE-Migraine
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00513681
Record Dates: First submitted 2025-10-28; First posted 2025-10-31 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Migraine; Chronic Migraine Headache; Refractory Migraine
Keywords: embolization; middle meningeal artery
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treatment (Experimental): Participants will undergo embolization of the middle meningeal arteries with Onyx.
  Interventions: Device: embolization of middle meningeal arteries

INTERVENTIONS:
Device: embolization of middle meningeal arteries — Participants will undergo embolization of the middle meningeal arteries with Onyx

SUMMARY:
This study is to test the safety and feasibility of a procedure called embolization of the middle meningeal arteries (MMA), using a product called Onyx. Embolization creates a plug in the arteries. MMA embolization with Onyx is not approved for use in patients with migraines, but is currently used in patients with subdural hematomas. The FDA is allowing the use of Onyx in this study. It is thought that by using Onyx to block the middle meningeal arteries, the amount of migraine-causing substances which are released into the brain's bloodstream will be reduced. The company that manufactures Onyx, Medtronic, is providing the supplies for this study.

Participants will be in the study for about 8 months after enrolling, including 6 months of follow up after the procedure. The participants will be asked to complete a daily headache diary and continue the participant's regular migraine medications. Participants will also have several clinic visits and be asked to provide blood samples for research.

ELIGIBILITY:
Inclusion criteria:

* Age 18<x<80
* Meets ICHD3 criteria for chronic migraine, (ICHD3, 1.3; with inclusion of ICHD3 1.1 and 1.2.1 only), with first migraine before age 50 (in concordance with previously published trials in migraine therapy36,39) . Patients must experience bilateral migraine symptoms.
* Satisfy criteria for refractory chronic migraine defined as failure of, inadequate response to, or inability to tolerate migraine preventatives in at least 2 classes. Migraine preventatives include beta-blockers, calcium channel blockers, anti-convulsants (valproic acid, topiramate), anti-depressants (venlafaxine, amitriptyline), CGRP monoclonal antibodies, botulinum toxin injections. Chronic migraines must have persisted for at least 12 months prior to enrollment and at least 6 months after failing 2 classes of medication.
* Has not used opiates or barbiturates as acute (rescue) therapy for migraine headache. Opiate or barbiturate use for reasons other than migraine is allowed. Other classes of acute migraine medications are acceptable. Acute (rescue, abortive) medications for migraines include acetaminophen, NSAIDs (ibuprofen, naproxen), gepants, triptans, anti-emetics (anti-nausea medications).
* Exclusion of secondary headache disorder which may cause migraines/symptoms, including MRI/MRA (performed as routine care showing no underlying lesion that may be causing headaches, within 3 years of screening).
* At least one migraine free day during the last month per headache diary.
* Minimum MIDAS score of 21 (reflecting severely disabling migraine, in concordance with ongoing MMA lidocaine infusion trial44).
* Able to read/write in English. Patients who are not English language users will not be enrolled as the study assessments are only validated in English.
* Able to sign informed consent for themselves.
* Able to complete study requirements/follow-up as outlined in study plan section 3.6.

Exclusion criteria:

* History of cranial or cervical vascular interventions or surgery, including craniotomy/craniectomy, shunt placement, stereoelectroencephalography, and carotid endarterectomy.
* A history of opiate or barbiturate use for the treatment of chronic migraine within one year.
* Current intracranial lesions as determined by routine care MRI for exclusion of secondary headache disorders.
* History of cranial radiation treatment.
* Patients with additional diagnoses under ICHD3 (such as hemiplegic migraine, basilar migraine, new daily persistent headache, or cluster headache) are ineligible
* Significant liver function impairment or serum creatinine > 2.0 mg/dL. Patients with elevated creatinine levels who are on dialysis may be eligible.
* History of systemic malignancy or auto-immune inflammatory disorders (such as multiple sclerosis, rheumatoid arthritis, autoimmune diseases).
* History of life-threatening allergy to radiographic contrast. Patients with this allergy may be eligible if it can be managed medically.
* Enrollment in another migraine study which could confound this study's endpoints, including undergoing any intervention or receiving an experimental drug under investigation for migraine therapy.
* Additional medical or social concerns which could confound this study's endpoints or otherwise create undue risk or interfere with the participant's ability to complete the study, as assessed by the PI.
* As this study is open only to patients with chronic migraine, which is refractory to treatment, patients who have previously been diagnosed with chronic migraine but now experience episodic migraine due to effective therapy are not eligible.
* Patients with additional diagnoses under ICHD3 (such as hemiplegic migraine, basilar migraine, new daily persistent headache, or cluster headache) are ineligible.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Number of specified adverse events related to the study | 30 days after procedure
  Strokes (ischemic and hemorrhagic), blindness, facial palsy, epidural hematoma, and death within 30 days of the embolization

CONTACTS AND LOCATIONS:
Overall Officials: Risheng Xu, MD, PhD, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No